CLINICAL TRIAL: NCT02999789
Title: Interventions to Help Asthma Clinical Adherence
Acronym: ITHACA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, San Francisco (Other)
Collaborators: Academic Pediatric Association (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 15-16445
Record Dates: First submitted 2016-12-16; First posted 2016-12-21 (Estimated); Results first posted 2023-04-18 (Actual); Last update posted 2023-04-18 (Actual); Status verified 2023-03

CONDITIONS: Asthma in Children; Humans; Hispanic Americans; Child
Keywords: Asthma/drug therapy; Medication Adherence/statistics & numerical data; Reminder Systems; Communication Barriers
MeSH Terms: conditions — Medication Adherence

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Intervention: Reminder System (Active Comparator): After an initial six week run-in period, participants will be randomized to either the intervention group or placebo group. The intervention group will have SMS reminder and audiovisual reminder functions turned on. SMS reminders will be sent twice daily to child's caregiver's cell phone reminding them to administer daily asthma medication. SmartInhaler with reminder function turned on that is attached to Inhaler medication will remind child's caregiver twice daily to administer daily asthma medication.
  Interventions: Device: SmartInhaler with reminder function turned on
- Placebo: Delayed Reminder System (Placebo Comparator): After an initial six week run-in period, participants will be randomized to either the intervention group or placebo group. The placebo group will have SMS reminder and audiovisual reminder functions turned off. The SmartInhaler will only function to measure daily adherence. Once intervention group has finished their 6 week period, this group will have intervention turned on.
  Interventions: Device: SmartInhaler

INTERVENTIONS:
Device: SmartInhaler with reminder function turned on — The SmartInhaler is a medication monitoring system that functions as a patient reminder device. It monitors asthma medication adherence and also functions by providing an audiovisual reminder.
  Arms: Intervention: Reminder System
Device: SmartInhaler — The SmartInhaler is a medication monitoring system manufactured by Adherium that also functions as a patient reminder device. It monitors asthma medication adherence and also functions by providing an audiovisual reminder.
  Arms: Placebo: Delayed Reminder System

SUMMARY:
To conduct a pilot test to estimate the effect of a novel reminder system in improving daily asthma controller medication adherence rates in children with monolingual Spanish-speaking guardians who have limited English Proficiency (LEP).

DETAILED DESCRIPTION:
The primary hypothesis is to conduct a pilot test to estimate the effect of the SmartInhaler device in improving daily asthma controller medication adherence rates in children with monolingual Spanish- speaking guardians who have LEP during a six-week intervention period when compared to baseline medication adherence rates in a preceding six-week run-in period. The secondary hypothesis is to determine whether the patient reminder system can improve asthma symptom control during the same six-week intervention period. The third hypothesis is to assess if there are specific, patient behavior characteristics which are associated with the success of a novel asthma medication reminder system.

ELIGIBILITY:
Inclusion Criteria:

1. The investigators will recruit 30 participants ages 5 to 17 years with a diagnosis of persistent asthma who require a daily inhaled corticosteroid metered dose inhaler and whose guardian is the person responsible for administering their daily asthma medication.
2. The investigators will recruit only participants who have received or receive care at San Francisco General Hospital's 6M Children's Health Center.
3. The investigators will recruit participants whose daily inhaled corticosteroid are metered dose inhalers (MDI) of either Flovent (fluticasone propionate) HFA (Hydrofluoroalkane) or Qvar (beclamethasone dipropionate) HFA.
4. The Investigators will recruit only participants whose guardian responsible for administering their daily asthma medication has Limited English Proficiency (LEP) and whose primary language is Spanish.

Exclusion Criteria:

1. The Investigators will exclude participants whose guardian responsible for administering their daily asthma medication does not have a Bluetooth enabled cell phone capable of receiving text messages.
2. The Investigators will exclude participants whose guardian responsible for administering their daily asthma medication does not have an available reliable power outlet where they can recharge the battery of their SmartInhaler.
3. The Investigators will exclude participants whose guardian responsible for administering their daily asthma medication is unable to demonstrate correct medication technique based on standard evaluation (Press, 2011) after completion of a standard teaching protocol.
4. The Investigators will exclude participants with chronic lung disease.
5. The Investigators will exclude participants who do not have an operating system of iOS or Android on their cell phone and who have no data plan with their cellular phone plan.
6. The Investigators will exclude participants whose asthma medication regimen is being managed by an asthma subspecialist or health provider outside of the 6M Children's Health Center at San Francisco General Hospital.
7. The Investigators will exclude participants who are using an inhaled long acting beta-agonist (LABA) as part of their asthma management plan.

Ages: 5 Years to 17 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 13 (Actual)
Dates: Start 2017-01; Primary Completion 2019-11 (Actual); Study Completion 2019-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Edward S Cruz, MD, MPH, Principal Investigator — University of California, San Francisco
Locations (1):
- Zuckerberg San Francisco General Hospital, San Francisco, California, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 13 participants were enrolled in total, 6 participants dropped out pre-randomization, and 4 participants were randomized to the intervention (reminder system) arm and 3 participants were randomized to the placebo (delayed reminder system) arm.
Period: Overall Study
Arm/Group | Intervention: Reminder System | Placebo: Delayed Reminder System
Started | 4 | 3
Completed | 3 | 0
Not Completed | 1 | 3
Not completed — Withdrawal by Subject | 0 | 1
Not completed — Became ineligible | 1 | 2

BASELINE CHARACTERISTICS:
Groups:
- Reminder System Arm Participants: After an initial six week run-in period, participants will be randomized to either the intervention group or placebo group. The intervention group will have SMS reminder and audiovisual reminder functions turned on. SMS reminders will be sent twice daily to child's caregiver's cell phone reminding them to administer daily asthma medication. SmartInhaler with reminder function turned on that is attached to Inhaler medication will remind child's caregiver twice daily to administer daily asthma medication.
  SmartInhaler with reminder function turned on: The SmartInhaler is a medication monitoring system that functions as a patient reminder device. It monitors asthma medication adherence and also functions by providing an audiovisual reminder.
- Delayed Reminder System Arm Participants: After an initial six week run-in period, participants will be randomized to either the intervention group or placebo group. The placebo group will have SMS reminder and audiovisual reminder functions turned off. The SmartInhaler will only function to measure daily adherence. Once intervention group has finished their 6 week period, this group will have intervention turned on.
  SmartInhaler: The SmartInhaler is a medication monitoring system manufactured by Adherium that also functions as a patient reminder device. It monitors asthma medication adherence and also functions by providing an audiovisual reminder.
- Enrolled But Not Randomized: Participants were enrolled but not randomized.
- Total: Total of all reporting groups
Arm/Group | Reminder System Arm Participants | Delayed Reminder System Arm Participants | Enrolled But Not Randomized | Total
Number analyzed (Participants) | 4 | 3 | 6 | 13
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 4 | 3 | 6 | 13
  Between 18 and 65 years | 0 | 0 | 0 | 0
  >=65 years | 0 | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 1 | 4 | 6
  Male | 3 | 2 | 2 | 7
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 4 | 3 | 6 | 13
  Not Hispanic or Latino | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 4 | 3 | 6 | 13

OUTCOME MEASURES:

1. Primary Outcome: Change in Percentage of Doses Received
Description: Medication adherence for each medication was calculated as a percentage of the total number of doses received during the study period divided by the total number of doses prescribed. As a result, this percentage ranged from 0 to 100. Medication adherence percentages during both the run-in and intervention periods were measured and the differences between doses received between the two time periods was calculated for each patient.
Time Frame: Baseline and 6 weeks post intervention
Measure: Median (Inter-Quartile Range); unit: Percentage of doses received
Arm/Group | Intervention: Reminder System | Placebo: Delayed Reminder System
Number analyzed (Participants) | 4 | 3
Percentage of doses received | 22.0 [7.5 to 91.4] | 12.4 [-34.9 to 60.7]

2. Secondary Outcome: Asthma Symptom Control Score Change
Description: The secondary hypothesis is to determine whether the patient reminder system can improve asthma symptom control during the same six-week intervention period. Asthma control will be measured by the Childhood asthma control test (C-ACT). The C-ACT is a 7 item scale, with scores ranging from 0 (poor asthma control) to 27 (complete asthma control). In general, a C-ACT score >19 indicates well-controlled asthma. Asthma symptom control scores during both the run-in and intervention periods were measured and the differences between scores between the two time periods was calculated for each patient.
Time Frame: Baseline and 6 weeks post intervention
Measure: Median (Inter-Quartile Range); unit: Score on a scale
Arm/Group | Intervention: Reminder System | Placebo: Delayed Reminder System
Number analyzed (Participants) | 4 | 3
Score on a scale | 3.0 [2 to 4] | 0 [-5 to 5]

3. Other Pre Specified Outcome: Type of Non-adherence
Description: The third hypothesis is to assess if there are specific, patient behavior characteristics which are associated with the success of a novel asthma medication reminder system. This will be assessed by the Reported Adherence to Medication survey (RAM)
Time Frame: Six weeks
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: Up to 18 weeks
Groups:
- Run-In Period (Placebo): During the Run-In period, we were measuring baseline adherence rates and no intervention was occurring.
- Intervention: Delayed Reminder System: After an initial six week run-in period, participants will be randomized to either the intervention group or placebo group. The placebo group will have SMS reminder and audiovisual reminder functions turned off. The SmartInhaler will only function to measure daily adherence. Once intervention group has finished their 6 week period, this group will have intervention turned on.
  SmartInhaler: The SmartInhaler is a medication monitoring system manufactured by Adherium that also functions as a patient reminder device. It monitors asthma medication adherence and also functions by providing an audiovisual reminder.
Arm/Group | Run-In Period (Placebo) | Intervention: Reminder System | Intervention: Delayed Reminder System
All-Cause Mortality (participants affected / at risk) | 0/13 | 0/4 | 0/3
Serious Adverse Events (participants affected / at risk) | 0/13 | 0/4 | 0/3
Other Adverse Events (participants affected / at risk) | 0/13 | 0/4 | 0/3

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol (2019-01-28): https://cdn.clinicaltrials.gov/large-docs/89/NCT02999789/Prot_000.pdf
  • Statistical Analysis Plan (2021-02-23): https://cdn.clinicaltrials.gov/large-docs/89/NCT02999789/SAP_001.pdf